CLINICAL TRIAL: NCT02514369
Title: Pharmacogenetics of New Antiretroviral Drugs
Brief Title: Pharmacogenomics of New Antiretrovirals
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: ARVLB01
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Some genetic polymorphisms are known to interfere with ARV metabolism and are therefore likely to explain some of the inter-individual variations (efficacy,toxicity,resistance) observed during ART. The most common form of human DNA variations consists of a change of a base in the nucleotide sequence of an individual at a given position, the single nucleotide polymorphism (SNP). Therefore,the purpose of this research will be the identification and characterization of the clinical impact of several SNPs in gene coding for transport proteins (e.g.ABCB1,ABCC1) and biotransformation enzymes (e.g.CYP3A4,CYP2B6) known to be involved in the pharmacokinetic pathway of selected ARV drugs for which the therapeutic response is difficult to predict. Aside,the influence of these SNPs on the response to treatment (CD4+cell,viral load) and on the toxicity will be evaluated. Plasma concentrations of ARV drugs correlate with therapeutic efficacy but also with the risk of toxicity and of virological failure, which is the basis of the therapeutic drug monitoring. However,given the intracellular location of HIV, analyzing intracellular drug concentrations is fundamental and the investigators will also focus of this new topic.

DETAILED DESCRIPTION:
Some genetic polymorphisms are known to interfere with ARV metabolism and are therefore likely to explain some of the inter-individual variations (efficacy,toxicity,resistance) observed during ART. The most common form of human DNA variations consists of a change of a base in the nucleotide sequence of an individual at a given position, the single nucleotide polymorphism (SNP). Therefore,the purpose of this research will be the identification and characterization of the clinical impact of several SNPs in gene coding for transport proteins (e.g.ABCB1,ABCC1) and biotransformation enzymes (e.g.CYP3A4,CYP2B6) known to be involved in the pharmacokinetic pathway of selected ARV drugs for which the therapeutic response is difficult to predict. Considering that CYP3A5 may represent up to 50% of the total hepatic CYP3A content in CYP3A5*1 allele carriers, the CYP3A5 genetic polymorphism may be therefore the most important genetic contributor not only to interindividual but also to interracial differences in CYP3A-dependent drug clearance.

Aside,the influence of these SNPs on the response to treatment (CD4+cell,viral load) and on the toxicity will be evaluated.

Plasma concentrations of ARV drugs correlate with therapeutic efficacy but also with the risk of toxicity and of virological failure, which is the basis of the therapeutic drug monitoring. However,given the intracellular location of HIV, analyzing intracellular drug concentrations is fundamental and the investigators will also focus of this new topic.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive treated with drug of interest

Exclusion Criteria:

* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV1-positive patients
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2012-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Impact of pharmacogenomics on plasma concentration of new antiretroviral drugs | up to 48 months
  The geometric mean (GM) of cell associated concentration and plasmatic concentration of ARV drug
Impact of pharmacogenomics on intracellular concentration of new antiretroviral drugs | up to 48 months
  The geometric mean (GM) of cell associated concentration and plasmatic concentration of ARV drug

CONTACTS AND LOCATIONS:
Overall Officials: Leila Belkhir, MD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Result] Belkhir L, De Laveleye M, Vandercam B, Zech F, Delongie KA, Capron A, Yombi J, Vincent A, Elens L, Haufroid V. Quantification of darunavir and etravirine in human peripheral blood mononuclear cells using high performance liquid chromatography tandem mass spectrometry (LC-MS/MS), clinical application in a cohort of 110 HIV-1 infected patients and evidence of a potential drug-drug interaction. Clin Biochem. 2016 May;49(7-8):580-6. doi: 10.1016/j.clinbiochem.2015.12.011. Epub 2015 Dec 29. PMID 26742721